CLINICAL TRIAL: NCT03545360
Title: Safety and Efficacy of the BTL-703 Treatment for the Non-invasive Lipolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-703-001
Record Dates: First submitted 2018-03-28; First posted 2018-06-04 (Actual); Last update posted 2018-06-04 (Actual); Status verified 2018-05

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): Treated group of subjects, serves as its own control
  Interventions: Device: BTL-703 (Treatment group)

INTERVENTIONS:
Device: BTL-703 (Treatment group) — Treatment with BTL-703 device

SUMMARY:
The study will evaluate safety and efficacy of the BTL-703 device for the non-invasive lipolysis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 22 years
* Voluntarily signed informed consent form

Exclusion Criteria:

* Implanted electronic device such as a cardiac pacemaker, bladder stimulator, spinal cord stimulator or electrodes for a myoelectric prosthesis, etc.
* Diabetics dependent on insulin or oral hypoglycemic medications
* Known cardiovascular disease such as arrhythmias, congestive heart failure
* Cardiac surgeries such as cardiac bypass, heart transplant surgery, pacemakers.
* Prior surgical interventions for body sculpting of thighs or buttocks such as liposuction
* Medical, physical or other contraindications for body sculpting/ weight loss
* Current use of medication known to affect weight levels and/or cause bloating or swelling and for which abstinence during the course of study participation is not safe or medically prudent
* Any medical condition known to affect weight levels and/or to cause bloating or swelling
* Active infection, wound or other external trauma to the area to be treated
* Pregnant, breast feeding, or planning pregnant before the end of the study
* Serious mental health illness
* Active or recurrent cancer or current chemotherapy and/or radiation treatment
* Negative affection to heat

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-01-01 (Estimated)

PRIMARY OUTCOMES:
Waist circumference reduction | 5 months
  The waist circumference measure will be conducted in accordance to the WHO STEPwise approach to surveillance (2008.) and NHLBI Obesity Education Initiative (2000.) recommendations. The waist circumference after the therapy will be compared to baseline.

SECONDARY OUTCOMES:
Serious adverse events following the treatment | 5 months
  Occurrence of serious adverse events will be followed throughout the whole study.
Photo evaluation | 5 months
  Correct identification of the pre- and post-treatment photos by blinded evaluators.
Subject Satisfaction | 5 months
  Subject Satisfaction Questionnaire will be given to subjects at every follow-up visit.
Therapy discomfort | 2 months
  Subject's discomfort (pain) level after each treatment will be assessed using the Discomfort Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Aesthe Clinic, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No